CLINICAL TRIAL: NCT01615536
Title: The Role of Canine Fossa Trephination in the Severely Diseased Maxillary Sinus
Acronym: CFT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: IWitterick (Other)
Responsible Party: Sponsor-Investigator, IWitterick, Otolaryngologist Head-Neck Surgeon, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Organization: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0211-A
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Disorder of Maxillary Sinus; Aspirin-sensitive Asthma With Nasal Polyps; Rhinosinusitis
Keywords: chronic rhinosinusitis; canine fossa trephine; canine fossa puncture
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canine fossa trephine group (CFT) (Experimental)
  Interventions: Procedure: Canine fossa trephine technique
- Non Canine fossa trephine group (NonCFT) (Active Comparator)
  Interventions: Procedure: Standard Endoscopic Sinus Surgery

INTERVENTIONS:
Procedure: Canine fossa trephine technique — Patients undergoing standard ESS and a canine fossa trephine technique, which is a 6 mm puncture in the anterior wall of the maxillary sinus, to allow standard sinus debrider blades and instruments to pass into the sinus to clear polyps in the maxillary sinus.
  Other Names: Canine fossa puncture
  Arms: Canine fossa trephine group (CFT)
Procedure: Standard Endoscopic Sinus Surgery — Patients undergoing standard ESS without canine fossa trephination with clearance of the maxillary sinus polyps via a wide maxillary antrostomy (WMA) with use of curved debrider surgical blades and instruments.
  Other Names: Functional Endoscopic Sinus Surgery
  Arms: Non Canine fossa trephine group (NonCFT)

SUMMARY:
The hypothesis of this study is that canine fossa trephination (CFT) improves surgical outcomes for patients with a severely diseased maxillary sinus.

DETAILED DESCRIPTION:
Chronic sinusitis (CRS) with nasal polyps and thick mucin in the sinuses adversely affects results from endoscopic sinus surgery (ESS) because failure to clear the disease leads to ongoing inflammation and symptoms. In particular a subset of CRS patients with thick eosinophilic mucin (EMCRS) develop recurrent symptoms and require further surgeries. ESS techniques for the maxillary sinus requires a WMA in the side wall of the sinus and the use of curved debrider instruments to clear the polyps. Sometimes this doesn't provide access to the inferior/floor and anterior/front aspects of the maxillary sinus due to the fact that the maxillary sinus is on the side of the nasal cavity at an angle. The CFT through the front wall of the sinus was developed years ago as an alternative approach to improve access to these areas. Both techniques are acceptable standard treatments and which one is initially used to address the maxillary sinus currently depends on surgeon preference. The role of CFT has been studied by Sathanatar et al (Laryngoscope 2005) and Lee et al (Laryngoscope 2008) which provided conflicting results. Differences in their study patients and methodology could explain the different outcomes. Hence this study is proposed to clarify the role of CFT in patients with extensive maxillary sinus disease to see whether initial use of CFT is more helpful than WMA in the severely diseased maxillary sinus with polyps and mucin. Findings from this study may improve surgical outcomes for CRS patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extensively opacified maxillary sinuses on CT scanning undergoing Endoscopic Sinus Surgery for Chronic Rhinosinusitis
* Patients with Eosinophilic Mucin Chronic Rhinosinusitis or fungal sinusitis disease undergoing Endoscopic Sinus Surgery for Chronic Rhinosinusitis
* Patients with Recalcitrant Chronic Rhinosinusitis undergoing Endoscopic Sinus Surgery for Chronic Rhinosinusitis
* Patients over the age of 18
* Patients able to give informed consent to participate in the study

Exclusion Criteria:

* Patients will be excluded if they are unable to undergo surgery due to co morbidities.
* Patients with previous Caldwell-Luc procedures
* Patients with pre existing paraesthesia of the upper teeth or gums
* Patients with destructive lesions of the maxilla
* Patients with systemic disease affecting the paranasal sinuses (e.g. Wegener's granulomatosis)
* Patients immune compromised

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Standard validated symptom scores | 6 months
  1. Chronic sinusitis survey
  2. SNOT (Sinonasal Outcome Test)22

SECONDARY OUTCOMES:
Ability to completely clear the maxillary sinus of all disease (e.g. polyps and eosinophilic mucus) | Measured during surgery
  Measured by using a surgeon survey
Surgical time spent clearing the maxillary sinus disease between the CFT and non-CFT groups | At the time of surgery
  Measured in minutes
Endoscopy scores | Measured at 2,6, 12 months
  1. Grade 0: Normal mucosa with no evidence of disease
  2. Grade 1: Edematous mucosa and/or eosinophilic mucus
  3. Grade 2: Polypoidal mucosa and/or eosinophilic mucus
  4. Grade 3: Polyps and fungal debris

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Witterick, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mt Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sathananthar S, Nagaonkar S, Paleri V, Le T, Robinson S, Wormald PJ. Canine fossa puncture and clearance of the maxillary sinus for the severely diseased maxillary sinus. Laryngoscope. 2005 Jun;115(6):1026-9. doi: 10.1097/01.MLG.0000162651.22019.4A. PMID 15933514
- [Background] Lee JY, Lee SH, Hong HS, Lee JD, Cho SH. Is the canine fossa puncture approach really necessary for the severely diseased maxillary sinus during endoscopic sinus surgery? Laryngoscope. 2008 Jun;118(6):1082-7. doi: 10.1097/MLG.0b013e318169028d. PMID 18388769
- [Background] Gliklich RE, Metson R. Techniques for outcomes research in chronic sinusitis. Laryngoscope. 1995 Apr;105(4 Pt 1):387-90. doi: 10.1288/00005537-199504000-00010. PMID 7715384
- [Background] Singhal D, Douglas R, Robinson S, Wormald PJ. The incidence of complications using new landmarks and a modified technique of canine fossa puncture. Am J Rhinol. 2007 May-Jun;21(3):316-9. doi: 10.2500/ajr.2007.21.3022. PMID 17621816
- [Background] Lund VJ, Mackay IS. Staging in rhinosinusitus. Rhinology. 1993 Dec;31(4):183-4. No abstract available. PMID 8140385